CLINICAL TRIAL: NCT04689711
Title: Generalizable Prognostic Models for Patient-Centered Decisions in COVID-19
Brief Title: Prognostic Models for COVID-19 Care
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: Northwell Health (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: PCORI-ME-1606-35555
Record Dates: First submitted 2020-11-20; First posted 2020-12-30 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Approximately 20% of patients hospitalized with COVID-19 require intensive care and possibly invasive mechanical ventilation (MV). Patient preferences with COVID-19 for MV may be different, because intubation for these patients is often prolonged (for several weeks), is administered in settings characterized by social isolation and is associated with very high average mortality rates. Supporting patients facing this decision requires providing an accurate forecast of their likely outcomes based on their individual characteristics.

The investigators therefore aim to:

1. Develop 3 CPMs in each of 2 hospital systems (i.e., 6 distinct models) to predict:

   i) the need for MV in patients hospitalized with COVID-19; ii) mortality in patients receiving MV; iii) length of stay in the ICU.
2. Evaluate the geographic and temporal transportability of these models and examine updating approaches.

   1. To evaluate geographic transportability, the investigators will apply the evaluation and updating framework developed (in the parent PCORI grant) to assess CPM validity and generalizability across the different datasets.
   2. To evaluate temporal transportability, the investigators will examine both the main effect of calendar time and also examine calendar time as an effect modifier.
3. Engage stakeholders to facilitate best use of these CPMs in the care of patients with COVID-19.

DETAILED DESCRIPTION:
There has been a proliferation of COVID-19 clinical prediction models (CPMs) reported in the literature across health systems, but the validity and potential generalizability of these models to other settings is unknown. Generally, most hospitals (and systems) do not have a sufficient number of cases (and outcomes) to develop models fit to their local population, and predictor variables are not uniformly and reliably obtained across systems. Therefore, pooling and harmonizing data resources and assessing generalizability across different sites is urgently needed to create tools that may help support decision making across settings. In addition, since best practices are rapidly evolving over time (e.g., proning, minimizing paralytics, lung-protective volumes, remdesivir, dexamethasone or other treatments), updating and recalibrating these CPMs is crucially important.

In the current PCORI Methods project, the investigators developed a CPM evaluation and updating framework including both conventional and novel performance measures. The investigators will use this framework to evaluate COVID-19 prognostic models in the largest cohort of COVID-19 patients examined to date, spanning 2 datasets from very different settings. As the COVID-19 pandemic affects different regions, with subsequent waves expected, identifying the most accurate, robust and generalizable prognostic tools is needed to guide patient-centered decision making across diverse populations and settings.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patient survivor
* Family member/caregiver of patient hospitalized for COVID-19
* Physician with experience caring for COVID-19 patients
* Other provider (pastoral care, nursing, respiratory therapy) with experience caring for COVID-19 patients

Exclusion Criteria:

* Not proficient in reading or speaking English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will include COVID-19 survivors; family members of COVID-19 patients; caregivers for COVID-19 patients; critical care physicians; palliative care physicians; hospitalists; nurses; respiratory therapists; leaders of our clinical ethics committees and pastoral care representatives.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in model discrimination (Model 1: need for MV in patients hospitalized with COVID-19) | 30 days from hospitalization
  Aim 1 Outcome: Changes in Area under receiver operating characteristic curve (AUC) [delta AUC] for models predicting the probability of: the need for MV in patients hospitalized with COVID-19.
Changes in model discrimination (Model 2: mortality in patients receiving MV) | 30 days from hospitalization
  Aim 1 Outcome: Changes in Area under receiver operating characteristic curve (AUC) [delta AUC] for models predicting the probability of: mortality in patients receiving MV.
Changes in model discrimination (Model 3: length of stay in the ICU) | 30 days from hospitalization
  Aim 1 Outcome: Changes in Area under receiver operating characteristic curve (AUC) [delta AUC] for models predicting the probability of: length of stay in the ICU.
Changes in model calibration (Model 1: need for MV in patients hospitalized with COVID-19) | 30 days from hospitalization
  Aim 1 Outcome-Changes in Harrell's E for models predicting the probability of: the need for MV in patients hospitalized with COVID-19.
Changes in model calibration (Model 2: mortality in patients receiving MV) | 30 days from hospitalization
  Aim 1 Outcome-Changes in Harrell's E for models predicting the probability of: mortality in patients receiving MV.
Changes in model calibration (Model 3: length of stay in the ICU) | 30 days from hospitalization
  Aim 1 Outcome-Changes in Harrell's E for models predicting the probability of: length of stay in the ICU.
Changes in net benefit (Model 1: need for MV in patients hospitalized with COVID-19) | 30 days from hospitalization
  Aim 1 Outcome-Changes in Net Benefit for models predicting the probability of: the need for MV in patients hospitalized with COVID-19.
Changes in net benefit (Model 2: mortality in patients receiving MV) | 30 days from hospitalization
  Aim 1 Outcome-Changes in Net Benefit for models predicting the probability of: mortality in patients receiving MV.
Changes in net benefit (Model 3: length of stay in the ICU) | 30 days from hospitalization
  Aim 1 Outcome-Changes in Net Benefit for models predicting the probability of: length of stay in the ICU.
Changes in model discrimination in external database after updating (Model 1: need for MV in patients hospitalized with COVID-19) | 30 days from hospitalization
  Aim 2 Outcome-Changes in Area under receiver operating characteristic curve (AUC) [delta AUC] for models predicting the probability of: the need for MV in patients hospitalized with COVID-19.
Changes in model discrimination in external database after updating (Model 2: mortality in patients receiving MV) | 30 days from hospitalization
  Aim 2 Outcome-Changes in Area under receiver operating characteristic curve (AUC) [delta AUC] for models predicting the probability of: mortality in patients receiving MV.
Changes in model discrimination in external database after updating (Model 3: length of stay in the ICU) | 30 days from hospitalization
  Aim 2 Outcome-Changes in Area under receiver operating characteristic curve (AUC) [delta AUC] for models predicting the probability of: length of stay in the ICU.
Changes in model calibration in external database after updating (Model 1: need for MV in patients hospitalized with COVID-19) | 30 days from hospitalization
  Aim 2 Outcome-Changes in Harrell's E for models predicting the probability of: the need for MV in patients hospitalized with COVID-19.
Changes in model calibration in external database after updating (Model 2: mortality in patients receiving MV) | 30 days from hospitalization
  Aim 2 Outcome-Changes in Harrell's E for models predicting the probability of: mortality in patients receiving MV.
Changes in model calibration in external database after updating (Model 3: length of stay in the ICU) | 30 days from hospitalization
  Aim 2 Outcome-Changes in Harrell's E for models predicting the probability of: length of stay in the ICU.
Changes in net benefit in external database after updating (Model 1: need for MV in patients hospitalized with COVID-19) | 30 days from hospitalization
  Aim 2 Outcome-Changes in Net Benefit for models predicting the probability of: the need for MV in patients hospitalized with COVID-19.
Changes in net benefit in external database after updating (Model 2: mortality in patients receiving MV) | 30 days from hospitalization
  Aim 2 Outcome-Changes in Net Benefit for models predicting the probability of: mortality in patients receiving MV.
Changes in net benefit in external database after updating (Model 3: length of stay in the ICU) | 30 days from hospitalization
  Aim 2 Outcome-Changes in Net Benefit for models predicting the probability of: length of stay in the ICU.

SECONDARY OUTCOMES:
Stakeholder perceptions, beliefs and opinions on COVID prediction models | 6 months
  Aim 3 Outcome-The outcome will be assessed with a codebook derived deductively from our structured interview guide to identify themes that emerge in the semi-structured sessions. Through focus groups held via synchronous video conferences, we will engage with patients and clinical providers to identify patient- and provider-reported themes that emerge in how clinical prediction models can support decision making in the care of patients with COVID-19. Themes will be identified through qualitative analysis of patient and provider feedback. We expect to elicit patient and provider beliefs, opinions and values around the scientific, ethical and pragmatic aspects of use of these models to support decision making.

CONTACTS AND LOCATIONS:
Overall Officials: David M Kent, MD, MS, Principal Investigator — Tufts Medical Center
Locations (2):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - Northwell Health (The Feinstein Institutes for Medical Research), Manhasset, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Clarification of Mortality Rate and Data in Abstract, Results, and Table 2. JAMA. 2020 May 26;323(20):2098. doi: 10.1001/jama.2020.7681. No abstract available. PMID 32330939
- [Background] Wynants L, Van Calster B, Collins GS, Riley RD, Heinze G, Schuit E, Bonten MMJ, Dahly DL, Damen JAA, Debray TPA, de Jong VMT, De Vos M, Dhiman P, Haller MC, Harhay MO, Henckaerts L, Heus P, Kammer M, Kreuzberger N, Lohmann A, Luijken K, Ma J, Martin GP, McLernon DJ, Andaur Navarro CL, Reitsma JB, Sergeant JC, Shi C, Skoetz N, Smits LJM, Snell KIE, Sperrin M, Spijker R, Steyerberg EW, Takada T, Tzoulaki I, van Kuijk SMJ, van Bussel B, van der Horst ICC, van Royen FS, Verbakel JY, Wallisch C, Wilkinson J, Wolff R, Hooft L, Moons KGM, van Smeden M. Prediction models for diagnosis and prognosis of covid-19: systematic review and critical appraisal. BMJ. 2020 Apr 7;369:m1328. doi: 10.1136/bmj.m1328. PMID 32265220
- [Background] Levy TJ, Richardson S, Coppa K, et al. Development and Validation of a Survival Calculator for Hospitalized Patients with COVID-19. medRxiv. 2020:2020.2004.2022.20075416.
- [Background] Tibshirani R. Regression Shrinkage and Selection via the Lasso. Journal of the Royal Statistical Society Series B (Methodological). 1996;58(1):267-288.
- [Background] Putter H, Fiocco M, Geskus RB. Tutorial in biostatistics: competing risks and multi-state models. Stat Med. 2007 May 20;26(11):2389-430. doi: 10.1002/sim.2712. PMID 17031868
- [Background] de Wreede LC, Fiocco M, Putter H. The mstate package for estimation and prediction in non- and semi-parametric multi-state and competing risks models. Comput Methods Programs Biomed. 2010 Sep;99(3):261-74. doi: 10.1016/j.cmpb.2010.01.001. Epub 2010 Mar 15. PMID 20227129
- [Background] van Klaveren D, Steyerberg EW, Gonen M, Vergouwe Y. The calibrated model-based concordance improved assessment of discriminative ability in patient clusters of limited sample size. Diagn Progn Res. 2019 Jun 6;3:11. doi: 10.1186/s41512-019-0055-8. eCollection 2019. PMID 31183411
- [Background] Jones AE, Trzeciak S, Kline JA. The Sequential Organ Failure Assessment score for predicting outcome in patients with severe sepsis and evidence of hypoperfusion at the time of emergency department presentation. Crit Care Med. 2009 May;37(5):1649-54. doi: 10.1097/CCM.0b013e31819def97. PMID 19325482
- [Background] Lim WS, van der Eerden MM, Laing R, Boersma WG, Karalus N, Town GI, Lewis SA, Macfarlane JT. Defining community acquired pneumonia severity on presentation to hospital: an international derivation and validation study. Thorax. 2003 May;58(5):377-82. doi: 10.1136/thorax.58.5.377. PMID 12728155
- [Background] Griffith GJ, Morris TT, Tudball MJ, Herbert A, Mancano G, Pike L, Sharp GC, Sterne J, Palmer TM, Davey Smith G, Tilling K, Zuccolo L, Davies NM, Hemani G. Collider bias undermines our understanding of COVID-19 disease risk and severity. Nat Commun. 2020 Nov 12;11(1):5749. doi: 10.1038/s41467-020-19478-2. PMID 33184277
- See also: Parent study funded through the Patient Centered Outcome Research Institute (PCORI) to develop evaluation and updating framework for clinical prediction models used in this study. — https://www.pcori.org/research-results/2016/understanding-and-improving-accuracy-clinical-prediction-models-heart-disease

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT04689711/Prot_SAP_000.pdf